CLINICAL TRIAL: NCT03099200
Title: UK HER2 Positive Breast Cancer Productivity & Utility Non-Interventional Study (PURPOSE)
Brief Title: An Observational Study Evaluating the Productivity and Health-Related Quality of Life of People With HER2 Positive Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML30098
Record Dates: First submitted 2017-03-31; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort 1: Participants with early breast cancer currently undergoing treatment (either chemotherapy and targeted HER2 therapy OR targeted HER2 therapy alone) will be observed.
  Interventions: Other: No Intervention
- Cohort 2: Participants with early breast cancer who have completed treatment and are in disease-free survival (i.e. no longer receiving loco-regional treatment, chemotherapy or targeted HER2 therapy; participants may still be receiving hormone therapy) will be observed.
  Interventions: Other: No Intervention
- Cohort 3: Participants receiving treatment for metastatic breast cancer will be observed.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention

SUMMARY:
The purpose of this study is to compare productivity (in terms of work or daily activity) and generic and disease-specific health-related quality of life of participants with HER2 positive early breast cancer currently receiving adjuvant treatment (with chemotherapy and/or targeted HER2 therapy), with participants who have completed adjuvant parenteral therapy, and participants with HER2 positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with early stage or metastatic (Stage IV) HER2-positive breast cancer (confirmed by the study site physician). [HER2-positive is defined as ImmunoHistoChemistry (IHC3+) and/or in situ hybridization (ISH) ≥2.0]
* Able to provide written, informed consent.
* Early Stage Breast Cancer (eBC) patients must have received at least 1 cycle of adjuvant anti-cancer therapy following surgery; metastatic breast cancer (mBC) patients must have received at least 1 cycle of treatment for their metastatic disease.

Exclusion Criteria:

* Unwilling or unable to consent.
* Unable to complete written quality of life questionnaires
* Partcipants with Eastern Cooperative Oncology Group (ECOG) Performance Status ≥3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with HER2 positive early breast cancer currently receiving adjuvant treatment (with chemotherapy and/or targeted HER2 therapy), or have completed treatment and in disease-free survival, or receiving treatment for metastatic breast cancer will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
A Comparison of Productivity, Assessed by Patient-Reported Work Productivity and Activity Impairment (WPAI) Questionnaire Score, of Participants in Cohort 1 vs Cohort 2 vs Cohort 3 | Baseline
  The WPAI is a patient-reported measure which assesses the effect of general health and symptom severity on work productivity and regular activities. The General Health questionnaire asks participants to estimate the number of hours missed from work due to reasons related and unrelated to their health problems, as well as the total number of hours worked in the preceding 7-day period. The percentage of participants reporting that they were employed (working for pay) was assessed at baseline along with absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), and activity Impairment. The score range for the scales of the WPAI is between 0 (no effect) to 100% (max effect).

SECONDARY OUTCOMES:
A Comparison of Generic Health Related Quality of Life (HRQoL), Assessed by EuroQoL Health Related Quality of Life - 5 Dimensions - 5 Levels (EQ-5D-5L) Score, of Participants in Cohort 1 vs Cohort 2 vs Cohort 3 | Baseline
  EQ-5D-5L is a standardized, participant-rated instrument for use as a measure of health outcomes. The EQ 5D-5L includes 2 components: the EQ-5D-5L descriptive system and the visual analogue scale (VAS). The EQ-5D-5L descriptive system provides a profile of the participant's health state in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each dimension, the participant is instructed to choose one of 5 levels that best describes their health on that day: "no problem" (1), "slight" (2), "moderate" (3), "severe" (4), or "unable/extreme" (5). The VAS is the participant's rating of their health on a scale of 0 "worst health you can imagine" to 100 "best health you can imagine".
A Comparison of Disease-Specific HRQoL, Assessed by Functional Assessment of Cancer Therapy-Breast (FACT-B) Score, of Participants in Cohort 1 vs Cohort 2 vs Cohort 3 | Baseline
  FACT-B was used as the breast cancer-specific quality-of-life measure. FACT-B consists of 5 subscale scores pertaining to 4 well-being dimensions (physical, social/family, emotional, functional) and additional breast cancer concerns. A total overall score is the sum of all subscales. Response options were 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- United Kingdom (14):
  - Nevill Hall Hospital, Abergavenny
  - Colchester General Hospital, Colchester, Essex
  - Royal Devon & Exeter Hospital; Oncology Centre, Exeter
  - Royal Surrey County Hospital, Guildford
  - Ipswich Hospital; Clinical Oncology, Ipswich
  - Barts and the London NHS Trust., London
  - St George's Hospital, London
  - Christie Hospital; Breast Cancer Research Office, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Mount Vernon Cancer Centre, Northwood
  - Nottingham City Hospital; Oncology, Nottingham
  - Royal Cornwall Hospital, Truro
  - Pinderfields General Hospital, Wakefield
  - Yeovil District Hospital; Macmillan Cancer Unit, Yeovil